CLINICAL TRIAL: NCT03140683
Title: Predictors of Scar Dehiscence in Patients With Previous Caesarean Section; a Study of Different Variables Tenderness Versus Non-stress Test
Brief Title: Predictors of Scar Dehiscence in Patients With Previous Caesarean Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: SDCS
Record Dates: First submitted 2017-05-03; First posted 2017-05-04 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cesarean Section; Dehiscence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: non-stress test — antepartum fetal monitoring

SUMMARY:
In recent decades, the percentage of Cesarean section deliveries has dramatically increased in most countries. Concomitantly, the rates of vaginal birth after Cesarean have decreased steadily.

The pregnant women with previous Cesarean section face a difficult choice for their next delivery between a trial of labor after Cesarean or repeat caesarean section delivery.

The performance of multiple Cesarean section exposes women to greater risks of complications; furthermore, the risk of complications increases with each subsequent Cesarean section.

In fact, women with previous Cesarean section are more likely to experience short and long-term maternal complications in future pregnancies, or a trial of labor after Cesarean, with the risk of [uterine dehiscence, uterine rupture, genitourinary tract damage, hemorrhage and hysterectomy, abnormal placentation (placenta previa and placenta accreta) and difficulties during surgery

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant full-term 37-42 weeks.
2. Previous one caesarean section

Exclusion Criteria:

1. Absolute indication of cesarean section in previous and in current pregnancy
2. Pregnant women with Hemoglobin <9
3. Pregnant women with bleeding tendency
4. Pregnant women with collagen disease
5. Pregnant women with pre-eclampsia and eclampsia
6. Pregnant women with gestational diabetes
7. Multiple pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study sample will be collected from Women's Health Hospital of Assiut University and Assuit Health Insurance Hospital
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
number of women with dehisensce scar and Non-stress test abnormalities | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No